CLINICAL TRIAL: NCT06301464
Title: Validation of Serum Pepsinogen II and Helicobacter Pylori Test in the Detection of Gastric Cancer in South Korea
Brief Title: Pepsinogen II and Helicobacter Pylori Test in Gastric Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, Seoul National University Bundang Hospital
Other Study IDs: B-2003-603-103
Record Dates: First submitted 2024-03-02; First posted 2024-03-08 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; Pepsinogen; Helicobacter pylori
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Serum pepsinogens and anti-H. pylori antibody
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with gastric neoplasms: Patients with gastric neoplasms
- Normal control: Normal control without gastric neoplasms

SUMMARY:
The aim of this study to validate the role of pepsinogens in gastric cancer screening.

DETAILED DESCRIPTION:
Serum pepsinogens (PGs) are the biomarkers for gastric cancer (GC), especially atrophic gastritis which is a precursor of intestinal type GC and severe gastric inflammation which is an indicator for diffuse type GC in young age. So, test for serum PGs can be used to identify high risk patients for GC. The aim of this study is to validate the role of PGs in GC screening.

Sera and the data from esophagogastroduodenoscopy and questionnaires are collected from study subjects, and PGs and anti-H. pylori (HP) antibody are measured. Area under the curve and receiver operating characteristic curve are calculated to identify the optimal cutoff values for PGs.

To validate the usefulness of PGs to predict risk of GC, the subjects are divided into two groups based on each cut-off value for each PG value. Adjusted odds ratios (ORs) and 95% CIs are calculated using multivariate logistic regression. Risk stratification is conducted by combining each PG value and anti-HP antibody in GC subtype.

ELIGIBILITY:
Inclusion Criteria:

* Who undergoes serum pepsinogens and anti-H. pylori antibody tests, and esophagogastroduodenoscopy during a health-screening examination at Seoul National University Hospital Gangnam center (SNUHGC) or Seoul National University Bundang Hospital (SNUBH)

Exclusion Criteria:

* Who do not receive serum pepsinogens or anti-H. pylori antibody studies
* Who do not receive esophagogastroduodenoscopy within 3 months before or after the date of serum pepsinogens and anti-H. pylori antibody tests
* Subjects with recent proton-pump inhibitor therapy 1 month prior to enrollment
* Subjects with prior history of gastrectomy
* Subjects with upper gastrointestinal neoplasms other than gastric adenoma/adenocarcinoma
* Subjects who do not agree to participate in the study or withdraw his/her consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who have undergone a blood test for serum pepsinogens and anti-H. pylori antibody, have undergone an esophagogastroduodenoscopy test three months before and after the blood test, have no other reason for exclusion, and have agreed to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 24000 (Estimated)
Dates: Start 2003-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The level of serum pepsinogens | At the time of enrollment
  To compare the level of serum pepsinogens between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Nayoung Kim, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No